CLINICAL TRIAL: NCT04923412
Title: Prospective Randomized Controlled Study on the Effects of Vagus Nerve Pulmonary Branch Preservation During Video-assisted Thoracic Surgery Lobectomy in Non-small Cell Lung Cancer: Can it Decrease Postoperative Cough and Pulmonary Complications
Brief Title: Vagus Nerve Preservation and Chronic Cough in Non-small Cell Lung Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kwhanmien Kim, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2007-625-007
Record Dates: First submitted 2021-05-23; First posted 2021-06-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Vagus Nerve Injuries; Cough
MeSH Terms: conditions — Lung Neoplasms; Vagus Nerve Injuries; Cough

STUDY DESIGN:
Intervention Model Description: 214 patients will be divided into two groups.
  1. Control group (N=107): Effort to preserve the pulmonary branch of vagus nerve preservation is not made in this group during mediastinal lymph node dissection
  2. Treatment group (N=107): Effort to preserve the pulmonary branch of vagus nerve preservation is made in this group during mediastinal lymph node dissection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary branch of vagus nerve preserved (Experimental): Pulmonary branch of vagus nerve is preserved during the mediastinal lymph node dissection using minimally invasive surgery
  Interventions: Procedure: Pulmonary branch of vagus nerve preserved
- Pulmonary branch of vagus nerve not-preserved (Experimental): Pulmonary branch of vagus nerve is not preserved during the mediastinal lymph node dissection using minimally invasive surgery
  Interventions: Procedure: Pulmonary branch of vagus nerve not preserved

INTERVENTIONS:
Procedure: Pulmonary branch of vagus nerve preserved — During the mediastinal lymph node dissection using minimally invasive surgery, efforts to preserve the pulmonary branch of vagus nerve is made.
  Arms: Pulmonary branch of vagus nerve preserved
Procedure: Pulmonary branch of vagus nerve not preserved — During the mediastinal lymph node dissection using minimally invasive surgery, efforts to preserve the pulmonary branch of vagus nerve is not made/ can be severed.
  Arms: Pulmonary branch of vagus nerve not-preserved

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide. Surgical resection is the main treatment for resectable non-small-cell lung cancer (NSCLC), and lobectomy with systemic mediastinal lymph node dissection is the standard surgical method. However, a significant number of patients experience postoperative chronic cough; it is observed in about 60% of patients during the first year of outpatient clinic follow-up, and persistently lasts in about 24.7-50% during the 5 year follow-up period.

Several studies showed the association between vagus nerve and chronic cough. The bronchopulmonary vagal afferent C-fibers are responsible for cough, chest tightness and reflex bronchoconstrictions. It is expected that during the mediastinal lymph node dissection, the inevitable injuries to the pulmonary branch of vagus nerve is largely responsible for development of chronic cough. In other words, preservation of pulmonary branch of vagus nerve may reduce the incidence of chronic cough and relevant detrimental effects on quality of life.

Therefore, this prospective, randomized and controlled clinical study, aims to evaluate the effect of vagus nerve preservation on postoperative chronic cough in patients undergoing lobectomy with mediastinal lymph node dissection. In addition, the feasibility and oncologic safety of preserving pulmonary branch of vagus nerve during mediastinal lymph node dissection with minimally invasive surgery compared with conventional mediastinal lymph node dissection with minimally invasive surgery will also be investigated.

This trial will provide a new basis for oncologically feasible, safe and effective new surgical technique for mediastinal lymph node dissection in patients with early lung cancer undergoing minimally invasive surgery. Furthermore, the preventive effect of vagus nerve preservation on incidence of chronic cough will be objectively be proven and thus help to broaden the current knowledge of the role of vagus nerve and postoperative chronic cough.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects clearly understand the purpose of the study, are willing and able to comply with the requirements to complete the study, and can sign the informed consent.
2. Clinically suspicious of non-small cell lung cancer or tissue confirmed preoperatively
3. Clinical stage T1-3/N0-1/M0
4. Preoperative ECOG performance status 0-1
5. Preoperative ASA class I-III
6. Preoperative pulmonary function test FEV1 ≥ 60%, DLCO ≥ 60%
7. Patients expected to achieve R0 (complete resection) via simple lobectomy and mediastinal lymph node dissection

Exclusion Criteria:

1. Patients who smoked within 2 weeks prior to operation
2. Patients who received antitussives and expectorants 2 weeks prior to operation
3. Patients who are pregnant or breast feeding
4. Patients with severe or uncontrolled psychological disorders
5. Patients with severe pulmonary adhesion
6. Patients who are ineligible for minimally invasive surgery; thoracotomy conversion
7. Patients diagnosed with other malignancies within 2 years prior to operation
8. Patients who received chemotherapy or radiotherapy within 6 months prior to operation
9. Patients suspicious of clinical N2 or received neoadjuvant therapy prior to operation
10. Patients with cough-related diseases; COPD, asthma, ILD, GERD
11. Patients suspicious of lymph node metastasis/invasion around vagus nerve during the preoperative clinical staging evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative measurement of postoperative cough | Preoperative day
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Qualitative measurement of postoperative cough | Postoperative day (discharge day, an average of 1 week)
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Qualitative measurement of postoperative cough | Postoperative 1 month follow up at outpatient clinic
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Qualitative measurement of postoperative cough | Postoperative 2 month follow up at outpatient clinic
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Qualitative measurement of postoperative cough | Postoperative 6 month follow up at outpatient clinic
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Qualitative measurement of postoperative cough | Postoperative 12 month follow up at outpatient clinic
  Cough Visual Analog Scale (VAS) will be used for survey. The Cough VAS is a numeric scale from 0-10 scale, with 0 indicating that patient experiences no distress from cough and 10 indicating severe distress from cough.
Quantitative measurement of postoperative cough | Preoperative day
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Quantitative measurement of postoperative cough | Postoperative day (discharge day, an average of 1 week)
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Quantitative measurement of postoperative cough | Postoperative 1 month follow up at outpatient clinic
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Quantitative measurement of postoperative cough | Postoperative 2 month follow up at outpatient clinic
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Quantitative measurement of postoperative cough | Postoperative 6 month follow up at outpatient clinic
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Quantitative measurement of postoperative cough | Postoperative 12 month follow up at outpatient clinic
  The Korean version of the Leicester Cough Questionnaire will be used for survey. Comparison of preoperative and and postoperative change in objective cough frequency and quality of life among patients using the Leicester Cough Questionnaire, which is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.

SECONDARY OUTCOMES:
Serum TRPA1, TRPV1, bradykinin, PGE2 measurements | Preoperative day
  Measurement of TRPA1 (ng/mL), TRPV1 (ng/mL), bradykinin (pg/mL), PGE2 (pg/mL) (released from C-fibers) via enzyme-linked immunosorbent assay (ELISA) test to quantitatively measure the injures of the vagus nerve during the mediastinal lymph node dissection.
Serum TRPA1, TRPV1, bradykinin, PGE2 measurements | Postoperative 1 day
  Measurement of TRPA1 (ng/mL), TRPV1 (ng/mL), bradykinin (pg/mL), PGE2 (pg/mL) (released from C-fibers) via enzyme-linked immunosorbent assay (ELISA) test to quantitatively measure the injures of the vagus nerve during the mediastinal lymph node dissection.
Serum TRPA1, TRPV1, bradykinin, PGE2 measurements | Postoperative 2 month follow up at outpatient clinic
  Measurement of TRPA1 (ng/mL), TRPV1 (ng/mL), bradykinin (pg/mL), PGE2 (pg/mL) (released from C-fibers) via enzyme-linked immunosorbent assay (ELISA) test to quantitatively measure the injures of the vagus nerve during the mediastinal lymph node dissection.
Pulmonary function test | Preoperative day
  Routine PFT (FEV1%, FEV1/FVC%) check to evaluate the effects of vagus nerve preservation in pulmonary function
Pulmonary function test | Postoperative 1 month follow up at outpatient clinic
  Routine PFT (FEV1%, FEV1/FVC%) check to evaluate the effects of vagus nerve preservation in pulmonary function
Pulmonary function test | Postoperative 2 month follow up at outpatient clinic
  Routine PFT (FEV1%, FEV1/FVC%) check to evaluate the effects of vagus nerve preservation in pulmonary function
Pulmonary function test | Postoperative 6 month follow up at outpatient clinic
  Routine PFT (FEV1%, FEV1/FVC%) check to evaluate the effects of vagus nerve preservation in pulmonary function
Pulmonary function test | Postoperative 12 month follow up at outpatient clinic
  Routine PFT (FEV1%, FEV1/FVC%) check to evaluate the effects of vagus nerve preservation in pulmonary function
Incidence of postoperative pulmonary complications, hospital stay and readmission, ICU care | from admission for operation to until the date of first documented postoperative complication or readmission, whichever came first), assessed up to 30 days
Histopathologic review of the total number of mediastinal lymph node dissected | through study completion, an average of 1 year
  Total number of dissected mediastinal lymph nodes and metastatic lymph nodes will be analyzed. Patient's preoperative clinical N stage and pathologic N stage will be compared; if pathologic N stage is higher than that of the clinical N stage, it will be considered as nodal upstaging.

CONTACTS AND LOCATIONS:
Overall Officials: Kwhanmien Kim, MD. PhD, Study Director — Department of Thoracic and Cardiovascular Surgery, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University, Seongnam-si, Bundang, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon JW, Moon JY, Kim SH, Song WJ, Kim MH, Kang MG, Lim KH, Lee SH, Lee SM, Lee JY, Kwon HS, Kim KM, Kim SH, Kim SH, Jeong JW, Kim CW, Cho SH, Lee BJ; Work Group for Chronic Cough, the Korean Academy of Asthma, Allergy and Clinical Immunology. Reliability and validity of a korean version of the leicester cough questionnaire. Allergy Asthma Immunol Res. 2015 May;7(3):230-3. doi: 10.4168/aair.2015.7.3.230. Epub 2014 Dec 18. PMID 25749761
- [Background] Al-Shamlan F, El-Hashim AZ. Bradykinin sensitizes the cough reflex via a B2 receptor dependent activation of TRPV1 and TRPA1 channels through metabolites of cyclooxygenase and 12-lipoxygenase. Respir Res. 2019 Jun 6;20(1):110. doi: 10.1186/s12931-019-1060-8. PMID 31170972
- [Background] Chen S, Huang S, Yu S, Han Z, Gao L, Shen Z, Kang M. The clinical value of a new method of functional lymph node dissection in video-assisted thoracic surgery right non-small cell lung cancer radical resection. J Thorac Dis. 2019 Feb;11(2):477-487. doi: 10.21037/jtd.2019.01.15. PMID 30962991
- [Background] Huang J, Luo Q, Tan Q, Lin H, Qian L, Ding Z. Evaluation of the surgical fat-filling procedure in the treatment of refractory cough after systematic mediastinal lymphadenectomy in patients with right lung cancer. J Surg Res. 2014 Apr;187(2):490-5. doi: 10.1016/j.jss.2013.10.062. Epub 2013 Nov 5. PMID 24300131
- [Background] Lin R, Che G. Risk factors of cough in non-small cell lung cancer patients after video-assisted thoracoscopic surgery. J Thorac Dis. 2018 Sep;10(9):5368-5375. doi: 10.21037/jtd.2018.08.54. PMID 30416784
- [Background] Liu Z, Liu Y, Xie C, Yang J, Zeng B, Yeung SJ, Cheng C. Vagus nerve and phrenic nerve guided systematic nodal dissection for lung cancer. J Thorac Dis. 2019 Sep;11(9):4021-4027. doi: 10.21037/jtd.2019.08.80. No abstract available. PMID 31656677
- [Background] Poghosyan H, Sheldon LK, Leveille SG, Cooley ME. Health-related quality of life after surgical treatment in patients with non-small cell lung cancer: a systematic review. Lung Cancer. 2013 Jul;81(1):11-26. doi: 10.1016/j.lungcan.2013.03.013. Epub 2013 Apr 4. PMID 23562675
- [Background] Sarna L, Evangelista L, Tashkin D, Padilla G, Holmes C, Brecht ML, Grannis F. Impact of respiratory symptoms and pulmonary function on quality of life of long-term survivors of non-small cell lung cancer. Chest. 2004 Feb;125(2):439-45. doi: 10.1378/chest.125.2.439. PMID 14769722
- [Background] Sawabata N, Maeda H, Takeda S, Inoue M, Koma M, Tokunaga T, Matsuda H. Persistent cough following pulmonary resection: observational and empiric study of possible causes. Ann Thorac Surg. 2005 Jan;79(1):289-93. doi: 10.1016/j.athoracsur.2004.06.045. PMID 15620960
- [Background] Spinou A, Birring SS. An update on measurement and monitoring of cough: what are the important study endpoints? J Thorac Dis. 2014 Oct;6(Suppl 7):S728-34. doi: 10.3978/j.issn.2072-1439.2014.10.08. PMID 25383207
- [Background] Watanabe A, Nakazawa J, Miyajima M, Harada R, Nakashima S, Mawatari T, Higami T. Thoracoscopic mediastinal lymph node dissection for lung cancer. Semin Thorac Cardiovasc Surg. 2012 Spring;24(1):68-73. doi: 10.1053/j.semtcvs.2012.03.002. PMID 22643666
- [Background] Yang P, Cheville AL, Wampfler JA, Garces YI, Jatoi A, Clark MM, Cassivi SD, Midthun DE, Marks RS, Aubry MC, Okuno SH, Williams BA, Nichols FC, Trastek VF, Sugimura H, Sarna L, Allen MS, Deschamps C, Sloan JA. Quality of life and symptom burden among long-term lung cancer survivors. J Thorac Oncol. 2012 Jan;7(1):64-70. doi: 10.1097/JTO.0b013e3182397b3e. PMID 22134070
- [Background] Zhu YF, Wu SB, Zhou MQ, Xie MR, Xiong R, Xu SB, Xu GW. Increased expression of TRPV1 in patients with acute or chronic cough after lung cancer surgery. Thorac Cancer. 2019 Apr;10(4):988-991. doi: 10.1111/1759-7714.13042. Epub 2019 Mar 18. PMID 30883022